

Title: A Dose-Ranging, Randomized, Parallel, Placebo-Controlled Study to Assess the Effect of TAK-954 on Gastrointestinal and Colonic Transit in Patients With Diabetic or Idiopathic Gastroparesis

NCT Number: NCT03281577

SAP Approve Date: 25 September 2018

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



## STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-954-2003

, applicable Terms of Use A Dose-Ranging, Randomized, Parallel, Placebo-Controlled Study to Assess the Effect of TAK-954 on Gastrointestinal and Colonic Transit in Patients with Diabetic or Idiopathic

Gastroparesis

Version: 1.0
Date: 25 September 2018

d by:

Prepared by:

rotocol Version: <Amendment 4>
Protocol Date: <11 September 2018>

Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

| 2.0 | | TABLE OF CONTENTS | |
|---|---|---|---|
| 1.0 | | TITLE PAGE | 1 |
| | 1.1 | Approval Signatures | 2 |
| 2.0 | | TABLE OF CONTENTS. | 1 7 |
| 3.0 | | LIST OF ABBREVIATIONS | 5 |
| 4.0 | | OBJECTIVES | |
| | 4.1 | Primary Objectives | _ |
| | 4.2 | OBJECTIVES Primary Objectives Secondary Objectives Additional Objectives | 7 |
| | 4.3 | Additional Objectives | 7 |
| | 4.4 | Study Design | 7 |
| 5.0 | | ANALYSIS ENDPOINTS | 9 |
| | 5.1 | Primary Endpoint | 9 |
| | 5.2 | Secondary Endpoints | 9 |
| | 5.3 | Safety Endpoints | 9 |
| | 5.4 | Exploratory Endpoints | 9 |
| 6.0 | | Additional Objectives Study Design ANALYSIS ENDPOINTS Primary Endpoint Secondary Endpoints Safety Endpoints Exploratory Endpoints DETERMINATION OF SAMPLE SIZE | 10 |
| 7.0 | | METHODS OF ANALYSIS AND PRESENTATION | 11 |
| , | 7.1 | General Principles | 11 |
| | | 7.1.1 Definition of Study Days and Study Visit Windows | 11 |
| | | 7.1.1 Definition of Study Days and Study Visit Windows 7.1.2 Missing Data Analysis Sets Dignosition of Suborts | 14 |
| , | 7.2 | Analysis Sets | 15 |
| , | 7.3 | Disposition of Subjects | 15 |
| , | 7.4 | Demographic and Other Baseline Characteristics | 15 |
| , | 7.5 | Medical History and Concurrent Medical Conditions | 15 |
| , | 7.6 | Medication History and Concomitant Medications | 16 |
| , | 7.7 | | 16 |
| , | 7.8 | Efficacy Analysis | 16 |
| | | 7.81 Primary Efficacy Endpoint(s) | 16 |
| | 0 | 7.8.2 Secondary Efficacy Endpoint(s) | 16 |
| 4 | | 7.8.3 Additional Efficacy Endpoint(s) | 16 |
| 0. | 7.9 | Pharmacokinetic/Pharmacodynamic Analysis | 17 |
| | | 7.9.1 Pharmacokinetic Analysis | 17 |
| | | 7.9.2 Pharmacodynamic Analysis | 17 |
| | | 7.9.2.1 Primary PD endpoint | 17 |
| | | 7.9.2.2 Secondary PD endpoint | 18 |

### 3.0 LIST OF ABBREVIATIONS

5HT4 serotonin

99mTc technetium-99m
111In indium chloride isotope

AC ascending
AE adverse event

ALT alanine aminotransferase
ANCOVA analysis of covariance
ANOVA analysis of variance
AST aspartate aminotransferase

AUC area under the concentration-time curve

 $AUC_{24}$  area under the concentration-time curve from time 0 to 24 hours

AUC<sub>24</sub>,ss area under the concentration-time curve from time 0 to time 24, at steady state

AUCτ area under the concentration-time curve during a dosing interval

AV atrioventricular
BP blood pressure
BMI body mass index
BUN blood urea nitrogen

%CV percent coefficient of variation

C<sub>max</sub> maximum observed concentration

C<sub>max,ss</sub> maximum observed concentration during a dosing interval, at steady state

C<sub>trough</sub> observed concentration at the end of a dosing interval

CPK creatine phosphokinase
CRF case report form
CYP cytochrome P450
DC Descending colon

eCRF electronic case report form

ECG electrocardiogram

EFI enteral feeding intolerance

FAS full analysis set

FDA Food and Drug Administration follicle-stimulating hormone

GC geometric center GCP Good Clinical Practice

GCSI Gastroparesis Cardinal Symptom Index

GGT  $\gamma$ -glutamyl transferase GI gastrointestinal

HbA1c glycosylated hemoglobin
HIV human immunodeficiency virus
hCG human chorionic gonadotropin

HR

**ICH** 

**ICU** 

**INR IRB** 

**IUD** 

ΙV

**IVRS** 

kcal

LFT(s) LDH LLN

**LOCF** 

MTD

MedDRA

**NOAEL NOEL** 

PD **PGx** 

PK PPS

patient-reported outcome PRO Pretreatment event PTE

QD Once daily QOL quality-of-life

corrected QT interval QTc

OT interval with Fridericia correction method QTcF

RS rectosigmoid colon serious adverse event SAE SAP statistical analysis plan **SDB** standard database

**SUSARs** suspected unexpected serious adverse reactions

supraventricular tachycardia

half-emptying time transverse colon

tables, listings, and graphs upper limit of normal Ventricular tachycardia

World Health Organization Drug Dictionary WHODrug

### 4.0 **OBJECTIVES**

### 4.1 **Primary Objectives**

To evaluate the dose-dependent effects of TAK-954 on gastric emptying time of solids in subjects with diabetic or idiopathic gastroparesis assessed by scintigraphy.

### 4.2 **Secondary Objectives**

- To evaluate the PD effects of TAK-954 on intestinal and colonic transit time assessed by scintigraphy To assess the safety and tolerability of multiple doses of TAK-954

  Additional Objectives

### 4.3



### Study Design 4.4

This is a phase 2a dose-ranging, randomized, parallel group, double-blind, placebo-controlled study evaluating the effects of TAK-954 on gastric, small bowel, and colonic transit in diabetic subjects reporting symptoms of gastroparesis with previously documented delay in stomach emptying or in subjects with diagnosis of idiopathic gastroparesis. Twelve subjects per treatment group will be evaluated.

This study consists of 3 periods and a Follow-up: a Screening Period, a Baseline Period (between Day -14 and Day -6), a Treatment Period (Days 1 to 4), and a Follow-up Phone Call (Days 10 to 14). Women of childbearing potential will receive an additional Follow-up Phone Call (Days 38-43).

Subjects will have an initial Screening Visit, then will undergo a baseline gastric emptying assessment with scintigraphy scans acquired at 0, 1, 2, 3, and 4 hours after radiolabeled meal, between Day -14 and Day -6 (Baseline Visit). At least 48 hours prior to baseline scintigraphy, female subjects must have a negative urine pregnancy test.

If eligibility criteria are fulfilled, subjects will be randomized on Day 1 to 1 of 4 treatment arms: TAK-954 0.1, 0.3, or 1 mg, or placebo. Subjects will receive TAK-954 or placebo as a 60-minute intravenous (IV) infusion (at any time in the morning prior to 12:00) once a day (QD) for 3 days starting on Day 1. Following the TAK-954 infusion on Day 2, subjects will undergo scintigraphic assessment of gastric, small bowel, and colonic transit of solids during the Treatment Period

The subjects will have pharmacokinetic (PK) samples collected as follows:

- Day 1: prior to dosing (0 hour) and at 0.5, 1 (end of infusion), 1.5, 2, and 4 hours after start of infusion.
- Day 2: prior to dosing (0 hour,), 0.5, 1 (end of infusion), 1.5, 2, 5, 7, and 9 hours after the start of the infusion.
- Day 3: prior to dosing (0 hour), 0.5, 1 (end of infusion), 1.5, and 2 hours after start of infusion, with an optional 4-hour sample.
- Day 4: 25 hours after the start of the infusion on Day 3 (48 hours after the administration of the radiolabeled meal on Day 2, same time as the 48-hour geometric center measurement).

During the study, subjects will complete a daily diary to record their bowel habits and as well as their global score using the GCSI. The On-Study Bowel Habit Diary Card will be dispensed at Screening to be completed daily from Screening and through the Treatment Period. The completed Bowel Habit Diary Card will be collected at the conclusion of the study.

All participating subjects will have a 6-hour Holter monitor placed at the Baseline Visit. On Day 1, subjects will have continuous ECG monitoring for up to 4 hours after the infusion, then continuous monitoring with a Holter monitor which will be placed prior to the first dose on Day 1 until the morning of Day 3.

Participants will undergo follow-up safety monitoring by phone 7-10 days post last treatment dose. The study will be considered completed after the last subject's Follow-up Phone Call.

### 5.0

### 5.1

The primary endpoint for this study is half-emptying time (T1/2) of gastric emptying of solids.

Secondary Endpoints

Colonic geometric center at 4 2.1

### 5.2

- Colonic filling at 6 hours (measure of small bowel transit time) after the radiolabeled meal.
- T1/2 of ascending colon emptying.
- The following PK parameters of TAK-954:
  - Area under the concentration-time curve during a dosing interval (AUCτ), Cmax, and observed concentration at the end of a dosing interval (Ctrough).

### 5.3 **Safety Endpoints**

- The percentage of subjects who experience at least 1 treatment-emergent adverse event.
- The percentage of subjects who discontinue due to an AE.
- The incidence of subjects who meet the markedly abnormal criteria for safety laboratory tests postdose.
- The incidence of subjects who meet the markedly abnormal criteria for vital sign measurements postdose.
- The percentage of subjects who meet the markedly abnormal criteria for safety 12-lead ECG parameters and Holter monitor postdose.

### 5.4 **Exploratory Endpoints**



PD

Table 5.a below summarizes data for the primary response measures and uses the percent coefficient of variation, (%CV) to estimate the effect size detectable with 80% power based on a 2 sample z-test (ie, assuming the variation values are known) at a 2-sided alpha level of 0.05. The effect size is the difference in group means as a percentage of the laboration. the laboratory, the sample size of 12 subjects per group provides 80% power to detect approximately 30% changes in the primary endpoints of the study: gastric emptying, and overall colonic transit. This magnitude of change is considered clinically significant. The ANCOVA should provide 80% power to detect similar (pairwise) differences using a pooled estimate of variation across all 3 groups and potentially even smaller effect sizes by adjusting for important covariates. The data from the scintigraphic transit studies are unpublished but based on the same methods proposed for this study.

**Summary of Detectable Effect Sizes for PD Endpoints** Table 6.a

| | Assuming n=12/Group in Each of the 4 Dose Groups | C | )<br>) | | |
|---|---|---|---|---|---|
| | Response Type | Mean | SD | %CV | Effect Size (%) † |
| | Gastric emptying of solids T1/2 min (n=319) | 122 | 29.8 | 24.5 | 34.2 |
| | Colonic filling at 6 h, % (n=63) | 44 | 29 | 66 | 79 |
| | GC at 24 h (n=220) | 2.4 | 0/9 | 36 | 52 |
| | Ascending colon T1/2 h (n=50) | 15.0 | 8.0 | 53 | 63 |
| o vo perti | Colonic filling at 6 h, % (n=63) GC at 24 h (n=220) Ascending colon T1/2 h (n=50) † Detectable with 80% power, α=0.05. | | | | |

### 7.0 METHODS OF ANALYSIS AND PRESENTATION

### 7.1 General Principles

Statistical analysis will be performed using the SAS System, Version 9.4.

Categorical data will be summarized as the number and percentage of subjects in each category. Continuous data will be summarized using descriptive statistics, including the number of subjects, mean, standard deviation (SD), median, minimum, and maximum. The coefficient of variation (%CV) and geometric mean will be included in the summary of continuous data where indicated.

Arithmetic means, geometric means, and medians will be presented to 1 more decimal place than the recorded data, and SDs will be presented to 2 more decimal places than the recorded data, where appropriate. Where applicable, confidence intervals about a parameter estimate will be presented using the same number of decimal places as the parameter estimate and p-values will be rounded to 3 decimal places prior to assessment of statistical significance.

All statistical tests and confidence intervals (CIs) will be 2-tailed at  $\alpha$ =0.05 level for significance unless otherwise stated. All study-related raw data for enfolled subjects, including derived data, will be presented in data listings.

## 7.1.1 Definition of Study Days and Study Visit Windows

Study Day 1 is defined as the date of the first dose of study drug. Other study days are defined relative to Study Day 1, with Day 1 being Study Day 1 and Day -1 being the day prior to Study Day 1. Study days prior to the first dose of study drug will be calculated as: [date of assessment/event – date of first dose of study drug]. Study days on or after the first dose of study drug will be calculated as: [date of assessment/event – date of first dose of study drug + 1]. Unless specified otherwise, for all PD, symptom assessment, and safety endpoints, baseline is defined as the last non-missing measurement prior to the first dose of study drug.

Scintigraphy will be performed at 0, 1, 2, 3, and 4 hours post-radiolabeled meal on baseline visit (Days -14 to Day -6); on Day 2 at every 0.5 hour for first 4 hours post radiolabeled meal, then hourly until 9 hours post start of infusion; on Day 3 at 1 hour post start of infusion; and on Day 4 at 25 hours post start of infusion on Day 3.

PK timepoints will be collected on Day 1 prior to dosing (0 hour) and at 0.5, 1, 1.5, 2, and 4 hours after start of infusion; on Day 2 prior to dosing (0 hour), 0.5, 1, 1.5, 2, 5, 7, and 9 hours after the start of the infusion; on Day 3 prior to dosing (0 hour), 0.5, 1, 1.5, and 2 hours after start of infusion, with an optional 4-hour sample; and on Day 4 at 25 hours post start of infusion on Day 3.

Vital signs will be collected upon arrival and departure from the Clinical Research and Trials Unit and at the time of the PK. Physical examination will be conducted prior to dosing on Days 1, 2, and 3. 12-lead ECG will be performed prior to each IV infusion, within 30 minutes post infusion, and at discharge on Days 1, 2, and 3; and at the Final Visit on Day 4 or Early

Termination Visit. In addition, a 12-lead ECG will be performed when needed, if a subject develops symptoms suggestive of cardiovascular origin (eg, dizziness, chest pain).

A schematic of the study design is included as Figure 7.a.

Figure 7.a **Schematic of study design** 







There will be no imputation of incomplete or missing data unless otherwise indicated.

Plasma concentrations that are below the limit of quantification (BLQ) will be treated as zero in the summarizing concentration values and deriving of PK parameters. These values will be flagged in the data listings.

### 7.2 Analysis Sets

The Full Analysis Set (FAS) will include all randomized subjects who receive at least 1 dose of study drug. Subjects in this set will be analyzed according to the treatment they were randomized to receive.

The per protocol set (PPS) analysis set is a subset of the FAS. The PPS consists of all subjects who do not violate the terms of the protocol in a way that would significantly impact the efficacy assessment. All decisions to exclude subjects from the PPS dataset will be made prior to the unblinding of the study and subject to clinical review. This analysis set will be for efficacy analyses only and can be considered as a sensitivity analysis in support of the primary analysis based on the FAS.

The Safety Analysis Set (SAF) will include all subjects who receive at least 1 dose of study drug. Subjects in this set will be analyzed according to the treatment that was actually received. Subjects in this analysis set will be used for demographic, baseline characteristics, and safety summaries.

The PK Analysis Set is defined as all subjects who receive at least 1 dose of study drug and have sufficient blood sampling to allow for PK evaluation.

### 7.3 Disposition of Subjects

A subject disposition summary will be provided. Subjects' study completion data, including reasons for premature termination, will be provided in listings and also summarized.

Significant protocol deviations will be summarized.

A summary of screening failures will also be provided.

### 7.4 Demographic and Other Baseline Characteristics

For continuous variables (age, weight, height, and body mass index [BMI]), summary statistics will be generated. BMI (in kg/m²) will be calculated using the subject's baseline height and weight measurements and summarized.

For categorical variables, the number and percentage of subjects in each category will be presented.

There will be no inferential analysis of demographic and baseline characteristics.

### 7.5 Medical History and Concurrent Medical Conditions

Medical history is defined as significant conditions or diseases that resolved at or prior to the time of informed consent. Concurrent medical conditions are defined as significant ongoing conditions or diseases that are present at signing of informed consent.

Medical history and concurrent medical conditions will be coded using the latest version of MedDRA, and will be summarized by treatment and overall using System Organ Class (SOC) and MedDRA preferred term (PT). The table will include number and percentages of subjects, and will be sorted in alphabetical order by SOC. Within an SOC, PTs are sorted in decreasing frequency based on the total number of subjects. A subject will only be counted once within a particular class even if he/she has multiple conditions/symptoms. Summaries will be based on the safety set. There will be no inferential analysis of medical history and concurrent medical conditions.

All medical history and concurrent medical condition data will be presented in data listing.

### 7.6 Medication History and Concomitant Medications

Medication history information to be obtained includes any medication relevant to eligibility criteria and efficacy/safety evaluation stopped at or within 48 hours prior to signing of informed consent. Medications used from signing of informed consent through the end of study will be considered as concomitant medications.

Medication history and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHODrug), and summarized by giving the number and percentage of subjects by preferred medication name within each therapeutic class, with therapeutic class sorted in alphabetical order and preferred term sorted in decreasing frequency based on the total number of subjects. If a subject report taking 2 drugs belonging to the same class, he/she will only be counted once within that class. Summaries of medication history and concomitant medication will be based on the safety set. There will be no inferential analysis of medication history and concomitant medications.

All medication history and concomitant medications data will be presented in data listing.

### 7.7 Study Drug Exposure and Compliance

The date and time of each dose for each subject will be reported in the data listing for all subjects. No summary statistics for the extent of exposure to study drug or compliance calculations will be performed for this study.

### 7.8 Efficacy Analysis

### 7.8.1 Primary Efficacy Endpoint(s)

Not applicable

### **7.8.2** Secondary Efficacy Endpoint(s)

Not applicable

### 7.8.3 Additional Efficacy Endpoint(s)

Not applicable

### 7.9 Pharmacokinetic/Pharmacodynamic Analysis

### 7.9.1 **Pharmacokinetic Analysis**

ms of Use PK parameters will be determined from the concentration-time data for all evaluable subjects. using non-compartmental analysis. Actual sampling times, rather than scheduled sampling times. will be used in all PK computations involving sampling times for plasma PK parameters.

For TAK-954, the following PK parameters including, but not limited to, will be calculated as appropriate:

- $AUC_{\tau}$ . Area under the concentration-time curve during a dosing interval (Day 1 to 3).
- C<sub>max</sub>: Maximum observed concentration (Day 1 to 3).
- C<sub>through</sub>: Observed concentration at the end of a dosing interval (Day 2 and 3).

The plasma concentration of TAK-954 will be summarized by treatment group over each scheduled sampling time point using descriptive statistics (N, arithmetic mean, SD, SE, CV%, median, minimum and maximum). In addition, the figures for mean plasma concentrations of TAK-954 versus time (linear and semi-log scale) will be generated, in overall population and by treatment group.

Additional plasma PK parameters may be calculated if necessary, in accordance with the Clinical Pharmacology Analysis Plan (CPAP).

### 7.9.2 Pharmacodynamic Analysis

The analyses and summaries for PD will be based on the FAS.

# 7.9.2.1 Primary PD endpoint

The primary PD endpoint is the half-emptying time (T1/2) of gastric emptying of solids.

Geometric mean of counts in anterior and posterior gastric regions of interest will be used to estimate by power exponential analysis, the proportionate emptying over time of counts from <sup>99m</sup>Tc solids and <sup>111</sup>In from the stomach. Gastric emptying from the power exponential analysis for the post injection period will be calculated and compared for the different treatments. The T<sub>1/2</sub> of gastric emptying of solids will be estimated by the linear interpolation using the slope of the 2 data points before and after 50% has emptied from the stomach. If less than 50% empty at 4 hours, the 3 data points at 180, 210, and 240 minutes will be used to project the time the  $T_{1/2}$ value.

Analysis of covariance (ANCOVA) methods will be used to assess the effect of treatment on the half-emptying time of gastric emptying of solids, including gastroparesis type (diabetic or idiopathic), age, gender, BMI, and the baseline measurement of gastric emptying  $T_{1/2}$  as covariates. Dunnett's test will be used to compare each treatment arm to placebo. Multiplicity adjusted and unadjusted 95% 2-sided confidence intervals will be presented. Normality will be tested using the Shapiro Wilk W test with criteria < 0.01. If normality is not achieved, a natural

Colonic geometric center at 4, 24, and 48 hours post meal will be estimated using geometric mean of counts in ascending, transverse, descending and rectosigmoid colon and stool (want) by factors of 1 to 5, respectively). The geometric center is the weighted and stool. At any time, the portion of weighting fact. weighting factors as follows:

$$(\%AC \times 1 + \%TC \times 2 + \%DC \times 3 + \%RS \times 4 + \%stool \times 5)/100 = geometric center$$

Thus, a high geometric center implies faster colonic transit. A geometric center of 1 implies that all isotope is in the ascending colon, and a geometric center of 5 implies that all isotope is in the stool.

Colonic filling at 6 hours post meal will be estimated by determining the amount of identified <sup>99m</sup>Tc -labeled solid meal within the colon at 6 hours with the value corrected for downscatter of radioactivity from the <sup>111</sup>Indium chloride isotope located within the same area appearing within the technetium window of analysis.

 $T_{1/2}$  of ascending colon emptying will be estimated by power exponential analysis of the proportionate emptying over time of counts from the colon. The primary data for this analysis will be the proportion of decay and depth-corrected counts in the ascending colon on the hourly scans on the first day of transit measurement and the 24 hour data. The  $T_{1/2}$  of ascending colon emptying is also estimated by plotting the activity-time curve for percent residing in the ascending colon; linear interpolation is used to connect points.

The effect of treatment on the secondary endpoints will also be assessed using an ANCOVA model. The covariates considered for inclusion in the analyses will be gastroparesis type (diabetic or idiopathic), age, gender, BMI, and the baseline measurement of the respective endpoint. Dunnett's test will be used to compare each treatment arm to placebo. Multiplicity adjusted and unadjusted 95% 2-sided confidence intervals will be presented. Normality will be tested using the Shapiro Wilk W test with criteria <0.01. If normality is not achieved, a natural log transformation may be done, and normality testing will be repeated. If normality is not achieved a non-parametric test (such as Kruskal Wallis) may be use.

### 7.10 Other Outcomes

Patient Reported Outcomes:

Information on the global score using the GCSI, as well as bowel movement frequency per day and average stool consistency on the Bristol stool form scale, will be tabulated by each day.

### 7.11 Safety Analysis

Safety analyses include adverse events (AEs), clinical laboratory parameters, vital sign parameters, 12-lead electrocardiogram (ECG) results.

All summaries of safety data are based on subjects in the Safety Set.

### 7.11.1 Adverse Events

All AE verbatim terms will be coded by SOC and PT using the latest version of MedDRA dictionary. SOCs will be sorted by alphabetical order. Within a SOC, PTs will be sorted in descending order based on the total number of subjects with AEs. For each category and overall, subjects reporting more than 1 occurrence for a term (SOC or PT) being summarized will be counted only once using the most extreme incident (most severe for the intensity tables and related for the relationship to study drug tables).

A treatment-emergent adverse event (TEAE) will be defined as an AE or serious adverse event (SAE) that started or worsened after first study drug administration and within 30 days of last dose of study drug (onset date – date of last dose +  $1 \le 30$ ). AEs with missing onset dates will be summarized with TEAEs regardless of severity and relationship to study medication.

TEAEs will be summarized by giving the number and percentage (N [%]) of subjects reporting any event for each term. The following is a list of TEAE summary tables to be generated.

- Overview of TEAEs (at both subject and event level).
- TEAEs by SOC and PT (at both subject and event level).
- Subject Mappings for TEAEs.
- TEAEs by SOC and PT by underlying disease condition (DG and IG).
- TEAEs by PT.
- Relationship of TEAEs to Study Drug by SOC and PT.
- Drug-Related TEAEs by SOC and PT.
- Intensity of TEAEs by SOC and PT.
- TEAEs leading to study discontinuation by SOC and PT.
- Treatment-emergent SAEs by SOC and PT.

An AE of Special Interest (serious or non-serious) is one of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator to Takeda may be appropriate.

### 7.11.2 Clinical Laboratory Evaluations

Clinical safety laboratory tests include hematology, serum chemistries, and urinalysis tests. Refer to Appendix A for the list of all clinical laboratory tests.

Descriptive statistics (N, mean, median, SD, minimum and maximum) of clinical safety laboratory variables will be summarized for baseline, postbaseline values, and change from baseline by treatment group and overall at each measurement. Only the scheduled measurements will be included in the summary. No inferential analysis will be performed.

Individual results for hematology laboratory tests and serum chemistry tests will be against the Takeda predefined laboratory marked.

Individual results for hematology laboratory tests and serum chemistry tests will be evaluated against the Takeda predefined laboratory markedly abnormal value (MAV) criteria (Appendix B). All subjects that meet the MAV criteria will be presented in a data listing. If a subject has a MAV for a particular laboratory test, all values for that subject and for that parameter will be listed. The number and percentage of subjects with at least 1 postbaseline markedly abnormal laboratory test result will be presented by treatment group and overall. All postbaseline clinical lab results within 7 days of the last dose, including scheduled and unscheduled measurements will be included in the MAV summaries. The mapping of the subjects with postbaseline results which meet the MAV criteria will be listed as a table.

All clinical laboratory data will be presented in both SI and conventional units in the data listings. Laboratory data outside of the normal reference range will be flagged on the listing along with values meeting MAV criteria.

### 7.11.3 Vital Signs

Vital sign measurements include body temperature, heart rate, respiratory rate, and blood pressure.

Descriptive statistics (N, mean, median, SD, minimum and maximum) of vital signs parameters will be summarized for baseline, postbaseline, and change from baseline at each scheduled time point. Only the vital signs collected at the scheduled visits or time points will be included in the summary. No inferential analysis will be performed.

All individual vital signs that meet Takeda's predefined criteria for markedly abnormal values (Appendix C) will be listed. The number and percentage of subjects with at least 1 postbaseline markedly abnormal vital sign measurement will be summarized. All postbaseline vital signs within 7 days of the last dose, including both scheduled and unscheduled measurements, will be included in the MAV summaries. The mapping of the subjects with postbaseline results which meet the MAV criteria will be listed as a table.

All vital sign data will be presented in the listings. Vital sign MAVs will be flagged in the listings.

### 7.11.4 12-Lead ECGs

The ECG parameters include heart rate, PR interval, QRS duration, QT interval, and QT interval with Fredericia's corrections (QTcF).

Descriptive statistics (N, mean, median, SD, minimum and maximum) of quantitative ECG data will be summarized for baseline, postbaseline, and change from baseline at each scheduled time point. Only the ECGs collected at the scheduled visits or time points will be included in the summary. No inferential analysis will be performed for the observed ECGs.

All individual ECGs that meet Takeda's predefined criteria for markedly abnormal values (Appendix D) will be listed. The number and percentage of subjects with at least one markedly abnormal ECG measurement will be summarized. All post dose ECGs within 7 days of the last dose, including both scheduled and unscheduled measurements will be summaries. The mapping of the subjects who

ect to the all All ECG and Holter monitor data will be presented in the listings. ECG MAVs will be flagged in the listings.

### 7.11.5 Other Observations Related to Safety

Not applicable

### 7.12 **Interim Analysis**

An interim analysis will be conducted when approximately half of the subjects have completed the study. Efficacy and safety data will be reviewed to determine if the study should be modified based on the interim analysis results. If needed, the changes will be related to dose selection, analysis E

analysis E

non-commercial use

Property of Takeda. For non-commercial use

Property of Takeda. sample size modification, or study termination.

# Changes in the Statistical Analysis Plan

Probeth of Takeda: For non-commercial use only and subject to the applicable Terms of Use

# Appendix A Clinical Laboratory Tests and Screening

### **Chemistry**

| Albumin | Alkaline phosphatase |
|---|---|
| ALT | AST |
| Blood urea nitrogen | Calcium |
| Bicarbonate | Chloride |
| Creatinine | Glucose |
| Gamma-glutamyl transferase | Sodium |
| Potassium | Bilirubin (total), if above ULN total bilirubin will be fractionated |
| Protein (total) | "K" |

## <u>Hematology</u>

| Erythrocytes (red blood cells [RBCs]) | Hemoglobin |
|---|---|
| Hematocrit | Platelets |
| Leukocytes (white blood cells [WBCs]) with absolute differential | 200 |

## <u>Urinalysis</u>

| · | |
|---|---|
| Protein | Glucose |
| Blood | Nitrite |
| Urine microscopy will b WBC/high-power field, | be performed if urinalysis is abnormal. Microscopy consists of RBC/high-power field, and casts. |
| rega: tot | ROLL |
| aroperty of Lan | |
| 6 tob | |

## Appendix B Criteria for Identification of Markedly Abnormal Laboratory Values

## Hematology—Criteria for Markedly Abnormal Values

| Parameter | Unit | Low Abnormal | High Abnormal |
|---|---|---|---|
| Hemoglobin | Both | <0.8 × LLN | >1.2 × ULN |
| Hematocrit | Both | <0.8 × LLN | >1.2 × ULN |
| RBC count | Both | <0.8 × LLN | >1.2 × ULN |
| WBC count | Both | <0.5 x LLN | >1.5 x ULN |
| Platelet count | Conventional | $<100 \text{ x } 10^3/\mu\text{L}$ | >450 x 10 <sup>3</sup> /μL |
| | SI | $<7100 x 10^9/L$ | >450 x 10 <sup>9</sup> /L |

LLN=lower limit of normal, RBC=red blood cell, ULN=upper limit of normal, WBC=white blood cell.

# <u>Serum Chemistry—Criteria for Markedly Abnormal Values</u>

| Parameter | Unit | Low Abnormal | High Abnormal |
|---|---|---|---|
| ALT | Both | 67 | >3x ULN |
| AST | Both | | >3x ULN |
| GGT | Both | ally are | >ULN - 2.5 x ULN if baseline was<br>normal; 2.0 - 2.5 x baseline if<br>baseline was abnormal |
| Alkaline phosphatase | Both | | >ULN - 2.5 x ULN if baseline was<br>normal; 2.0 - 2.5 x baseline if<br>baseline was abnormal |
| Total bilirubin | Conventional | | >ULN - 1.5 x ULN if baseline was normal; > 1.0 - 1.5 x baseline if baseline was abnormal |
| | COM | | >ULN - 1.5 x ULN if baseline was<br>normal; > 1.0 - 1.5 x baseline if<br>baseline was abnormal |
| Albumin | Conventional | <3 g/dL | |
| | SI | <30 g/L | |
| Total protein | Both | <0.8x LLN | >1.2x ULN |
| Creatinine | Conventional | | >2.0 mg/dL |
| 79. | SI | | >177 μmol/L |
| Blood urea nitrogen | Conventional | | >30 mg/dL |
| 12/ | SI | | >10.7 mmol/L |
| Sodium | Conventional | <130 mEq/L | >150 mEq/L |
| 0 | SI | <130 mmol/L | >150 mmol/L |
| Potassium | Conventional | <3.0 mEq/L | >5.5 mEq/L |
| • | SI | <3.0 mmol/L | >5.5 mmol/L |
| Glucose | Conventional | <55 mg/dL | >180 mg/dL |
| | SI | <3 mmol/L | >10 mmol/L* |
| Chloride | Conventional | <75 mEq/L | >126 mEq/L |
| | SI | <75 mmol/L | >126 mmol/L |

| | Parameter | Unit | Low Abnormal | High Abnormal |
|---|---|---|---|---|
| | Calcium (corrected) | Conventional | Corrected serum calcium<br>of <lln -="" 8.0="" dl;<br="" mg=""><lln -="" 2.0="" l;<br="" mmol="">Ionized calcium <lln -<br="">1.0 mmol/L</lln></lln></lln> | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; Ionized calcium >ULN - 1.5 mmol/L |
| | | SI | Corrected serum calcium of <lln -="" 1.0="" 2.0="" 8.0="" <lln="" calcium="" dl;="" ionized="" l;="" l<="" mg="" mmol="" td=""><td>Ionized calcium &gt;ULN - 1.5 mmol/L</td></lln> | Ionized calcium >ULN - 1.5 mmol/L |
| | Bicarbonate | Conventional | <8.0 mEq/L | |
| - | ALT=alanine aminotransfe<br>normal, ULN=upper limit of<br>Unless for patients wh | SI brase, AST=aspartate a of normal. o have Diabetic at base | <8.0 mmol/L<br>aminotransferase, GGT=γ-gluta<br>seline. | amyl transferase, LLN=lower limit of |
| | akedai. For n | on commercia | <8.0 mmol/L aminotransferase, GGT=γ-gluta seline. | |
| Property | of Takedai. For | | | |

# Appendix C Criteria for Abnormal Changes from Baseline of Vital Signs

| 11 | | , | 0 | |
|---|---|---|---|---|
| Parameter | Unit | Lower Criteria | Upper Criteria | |
| Heart Rate | bpm | <60 | >120 | nin. |
| Systolic blood pressure | mm Hg | <90 | >140 | |
| Diastolic blood pressure | mm Hg | <60 | | |
| Body temperature | °C | <35.6 | >37.7 | |
| | °F | <96.1 | >99.9 | |
| | | | 200 | |
| Body temperature Body temperature | | | *Ke | |
| | | | 60 | |
| | | : 00 | | |
| | | IOI | | |
| | | 720 | | |
| | | Sille | | |
| | | KI | | |
| | 0 | 0, | | |
| | JSE | ) | | |
| | o C | | | |
| | airie | | | |
| | COL | | | |
| | 1,00 | | | |
| , 100 | | | | |
| ₹0, | | | | |
| · | | | | |
| 1600 | | | | |
| 1 St | | | | |
| 4 | | | | |

# Appendix D Criteria for Markedly Abnormal Values for the 12-Lead ECG Parameters

| | 1 1 | V | |
|---|---|---|---|
| | Parameter | Lower Criteria | Upper Criteria |
| | Heart rate | <50 beats per minute | >120 beats per minute |
| | PR | ≤120 milliseconds | ≥200 milliseconds |
| | | | >500 milliseconds OR |
| | QTcF Interval | | ≥500 milliseconds <u>OR</u> |
| | | | ≥30 milliseconds change from baseline <u>and</u> ≥450 milliseconds |
| | QRS | ≤60 milliseconds | ≥120 milliseconds |
| Properto | of takeda. For no | ≤60 milliseconds Share only and share only and sh | Subject to the |

# ELECTRONIC SIGNATURES

| | | Server Date |
|---|---|---|
| Signed by | Meaning of Signature | (dd-MMM-yyyy HH:mm 'UTC') |
| PPD | Biostatistics Approval | (dd-MMM-yyyy HH;mm 'UTC')<br>25-Sep-2018 19:52 UTC |
| | Statistical Approval | 26-Sep-2018 <b>02:02</b> UTC |
| | Clinical Pharmacology Approval | 26-Sep-2018 15:24 UTC |
| | Pharmacovigilance Approval | 27-Sep-2018 11:46 UTC |
| | Clinical Science Approval | 28-Sep-2018 08:10 UTC |
| Property of Takeda. For non-con | nnercial use only and sur | |